CLINICAL TRIAL: NCT00273078
Title: Experimental Study About Tongue Interactions With Teeth and Palate During Speech, Using Strain Gauge Transducer and Complete Denture. Comparison of Adaptation Phenomenon's Between Patients With New Complete Denture.
Brief Title: Tongue Pressure Recording During Speech
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Other Study IDs: 2005.390
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Complete Toothless
Keywords: Speech,; tongue,; pressure,; transducer,; complete denture
MeSH Terms: conditions — Speech

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This research is about tongue's pressure during speech, using a complete denture which allows respecting tongue and speech physiology at the best.

A strain gauge transducer is placed inside this prosthodontics device. During speech, the pressure and the sounds are recording. The analysis of the twos signals should explain what pressure is needed for what sound. The comparison between old complete denture wearers and new one is realized to provide informations about tongue adaptation's phenomenon.

ELIGIBILITY:
Inclusion Criteria:

new prosthodontics device or change of prosthodontics device male or female Age upper 18 French as native language

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte GROGOGEAT, md, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Brigitte GROGOGEAT, Lyon, France